CLINICAL TRIAL: NCT03393117
Title: Prospective, Randomized, Blinded Comparison of Bupivacaine Versus Liposomal Bupivacaine For Breast Pain Management After Unilateral, Immediate Breast Reconstruction
Brief Title: Bupivacaine Versus Liposomal Bupivacaine For Breast Pain Management After Breast Recontruction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE10117
Record Dates: First submitted 2017-12-26; First posted 2018-01-08 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Reconstruction; Bupivacaine; Liposomal Bupivacaine
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine; Narcotics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Medication utilized will be blinded in the chart per inpatient pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine + Bupivacaine (Experimental): This group will receive a long-acting pain medicine, Liposomal Bupivacaine, injected into the breast muscles during surgery. All patients will receive patient-controlled analgesia pump and oral narcotics as indicated post surgery.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Bupivacaine; Drug: Patient-Controlled Analgesia Pump; Drug: Oral Narcotic
- Bupivacaine (Active Comparator): This group will receive the same pain medication, Bupivacaine, but in the standard formulation, injected into the breast muscles during surgery. All patients will receive patient-controlled analgesia pump and oral narcotics as indicated post surgery.
  Interventions: Drug: Bupivacaine; Drug: Patient-Controlled Analgesia Pump; Drug: Oral Narcotic

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 20mL vial of Liposomal Bupivacaine (266 mg). The infiltration technique for Liposomal Bupivacaine will be 80mL injected into either hemi-abdomen as a transversus abdominous plane (TAP) block via ultrasound guidance. The other 80mL will be utilized in the operative breast for the field blocks (20mL), pectoralis 1 (20mL), pectoralis 2 (20mL) and serratus anterior (20mL) blocks.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine + Bupivacaine
Drug: Bupivacaine — 20mL vial of 0.25% Bupivacaine. The field blocks (20mL), pectoralis 1 (20mL), pectoralis 2 (20mL) and serratus anterior (20mL) blocks will be performed with 0.25% Bupivacaine.
  Other Names: Sensorcaine-Methyl Paraben Free (MPF) Spinal; Sensorcaine-MPF; Sensorcaine; ReadySharp Bupivacaine; P-Care M; Marcaine Spinal; Marcaine Preservative Free; Marcaine; Bupivacaine Spinal
Drug: Patient-Controlled Analgesia Pump — The patient-controlled anesthesia will be filled with morphine or hydromorphone. Pumps will be programmed be on demand only with no basal rate.
  Other Names: intravenous narcotic
Drug: Oral Narcotic — Oral narcotics will be offered when the patient's diet is advanced as tolerated, typically post-operative day 1.

SUMMARY:
The purpose of this study is to determine the most effective way to control post-operative breast pain for patients undergoing a unilateral, immediate breast reconstruction.

DETAILED DESCRIPTION:
This is a randomized controlled study to compare the effectiveness of a breast nerve block performed with bupivacaine as compared to liposomal bupivacaine in providing postsurgical analgesia in patients undergoing unilateral abdominally-based breast reconstruction at time of mastectomy.

OBJECTIVES

1. Compare the amount of postoperative narcotic use in patients receiving a bupivacaine or liposomal bupivacaine pectoralis and serratus anterior nerve block. Compare these groups to a retrospective control cohort who received local anesthetic infusion but did not receive any nerve block.
2. Examine the incidence of narcotic-related side effects in the experimental groups by documenting incidents of nausea and vomiting, time to first ambulation, liquid and solid oral intake.
3. Survey patient satisfaction with pain management using a visual analog scale during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have a unilateral, immediate breast reconstruction

Exclusion Criteria:

* Pregnant
* Concurrent or recent medical condition that could interfere with study participation including:

  * Hepatitis
  * Alcohol/substance abuse
  * Uncontrolled psychiatric disorders
  * Known allergy
  * Contraindication to amide-type local anesthetics, opioids, or propofol.
* Body weight of less than 50 kg
* Participated in another study involving an investigational medication within the prior 30 days
* Taking analgesics (i.e., nonsteroidal anti-inflammatory drugs, acetaminophen, or opioids), antidepressants, or glucocorticoids within the 3 days before surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
total post-operative narcotic utilization | Up to 72 hours post-operative
  post-operative pain as measured by total post-operative narcotic utilization standardized to milligrams of morphine.

SECONDARY OUTCOMES:
at rest pain score on visual analog scale | Up to 72 hours post-operative
  0-100 score of self-reported pain
coughing pain score on visual analog scale | Up to 72 hours post-operative
  0-100 score of self-reported pain
number of incidents of nausea reported by patient | Up to 72 hours post-operative
  self-report of nausea
number of incidents of vomiting reported by patient | Up to 72 hours post-operative
  number of times a patient vomits
time to first ambulation | Up to 72 hours post-operative
time to first liquid intake | Up to 72 hours post-operative
time to first solid intake | Up to 72 hours post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Risal Djohan, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center